CLINICAL TRIAL: NCT02785302
Title: CATCH: Comprehensive Assessment of Transition and Coordination for HIV-Positive Youth as They Move From Adolescent to Adult Care
Brief Title: Transitioning HIV+ Adolescents to Adult Care: Exploring Adolescent and Adult Medicine Clinics Role in the Process
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 135
Record Dates: First submitted 2015-10-19; First posted 2016-05-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-12

CONDITIONS: HIV
Keywords: Pediatric; HIV; Transition; Adult Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents and Young Adults:: Behaviorally-infected, HIV-positive, adolescents and young adults enrolled in ATN 125, aged 18 through 24, inclusive who are transition eligible. All subjects with available endpoint data will be included in the analysis.
- AMTU and Adult Clinic Staff: Clinical staff at the Adolescent Medical Trials Units (AMTUs) and at adult clinics where the AMTUs refer their transitioning patients will be recruited to complete quantitative surveys and semi-structured interviews.

SUMMARY:
This is a multi-site, longitudinal study and it describes the transition process of behaviorally-infected HIV-positive youth as they move from pediatric- and adolescent-specific care to adult care. To achieve this goal, the transition process is characterized from the perspectives of HIV-positive youth, Adolescent Medicine Trials Unit (AMTU) clinic staff, and receiving adult clinic staff.

DETAILED DESCRIPTION:
The changes associated with transition to adult clinical care may increase the likelihood that an adolescent will drop out of care, which results in poorer outcomes. Disengagement from care has implications for health. Disruption in medication can increase viral load (VL), and intensify the potential for co-morbidities and transmission efficiency . Thus, successful transition to adult care is especially important for HIV-positive adolescents (compared to other chronic diseases) as they will need to maintain clinic visits and medication adherence across their lifespan to remain healthy and maintain a low VL to reduce the potential for transmission in the context of other developmental and psychosocial changes and challenges. The ultimate goal of this study is to represent the key places - youth, adolescent clinic and adult clinic - where transition interventions could be targeted and to collect data to capture the key elements and modifiable variables at each level. This study will contribute to existing research by providing transition research on HIV, which differs from other congenital or acquired chronic conditions due to it being an infectious disease; by prospectively following youth as they transition; and by providing transition research from the perspective of receiving adult clinics. It will also illustrate how each level- youth, adolescent clinic and adult clinic - is situated within a specific context and how these levels interact to affect transition outcomes.

This is a multi-method, longitudinal design research study. Subjects must be enrolled in ATN 125 at the time of the ATN 135 baseline visit. There will be no randomization procedures. During the 39-week study, surveys will be administered to adolescents and young adults transitioning to adult care via Audio Computer Assisted Self Interviews (ACASIs), which will collect data on individual (e.g., psychosocial and behavioral) and clinical factors affecting transition at 0 and 39 weeks. Demographic, biomedical, antiretroviral therapy (ART) and healthcare utilization visit information collected through ATN 125 medical chart abstraction will also become part of the ATN 135 subject dataset. One-time phone surveys and interviews with AMTU and adult clinic staff will also be conducted to collect information on transition protocols as well as review of any documentation of existing transition protocols (e.g., transitioning SOP). Outcome measures will include pre- and post-transition VL and other measures of physical and psychosocial health status to compare individuals with different patterns and outcomes of transition.

ELIGIBILITY:
Adolescents and young adults

Inclusion Criteria

To be considered eligible to participate in 135, behaviorally-infected HIV-positive adolescents and young adults must be:

* Enrolled in ATN 125
* Be transition eligible. Transition eligible means that the youth are either (a) age 18 through 24 years old and planning to transition to adult medical care within six months after ATN 135 enrollment or (b) 24 years old and not actively planning to transition to adult medical care.
* Willing and able to provide consent to participate.

Exclusion Criteria

To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to provide true informed consent or participate in the baseline ACASI;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior) at the time of consent or the baseline ACASI;
* At the time of consent, intoxicated or under the influence of alcohol or other substances to such an extent that in the opinion of the study staff, the ability to give true informed consent is impaired; or
* At the time of the baseline ACASI, intoxicated or under the influence of alcohol or other substances to such an extent that in the opinion of the study staff, the subject's ability to understand and answer the questions may be impaired and negatively impact the integrity of the research data.

AMTU and Partner Adult Clinic Staff

To be considered eligible to complete the AMTU and partner adult clinic surveys and semi-structured interviews, an individual must meet all of the criteria listed below.

* Being a clinical staff (e.g., healthcare providers, social workers, case managers, transition person) at either an AMTU or AMTU-affiliated site or partner adult clinic;
* Supporting (in any capacity) transition efforts for HIV-positive adolescents; and
* Willing and able to provide verbal consent for surveys and semi-structured interviews.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Behaviorally-infected HIV-positive adolescents and young adults between the ages of 18 and 24 years, are recruited to complete computer assisted interviews to characterize the transition process and outcomes.
  AMTU staff and partner adult clinic staff are recruited to complete quantitative surveys and semi-structured interviews over the phone to explore transition processes and protocols. There are no minimum or maximum age criteria that staff must meet .
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Transition Expectations and Experiences as assessed by the ACASI (comparison between pre- and post-transition) | Baseline
Transition Expectations and Experiences as assessed by the ACASI (comparison between pre- and post-transition) | 39 weeks
Patterns of Transition as assessed by the ACASI, as well as medical and appointment records abstraction (comparison between pre- and post-transition) | Baseline
Patterns of Transition as assessed by the ACASI, as well as medical and appointment records abstraction (comparison between pre- and post-transition) | 39 weeks
Patterns of Engagement in Care as assessed by the ACASI, as well as medical and appointment records abstraction (assessment over time from point of transition) | Baseline
Patterns of Engagement in Care as assessed by the ACASI, as well as medical and appointment records abstraction (assessment over time from point of transition) | 39 weeks

SECONDARY OUTCOMES:
Transition Protocols at AMTUs and Adult Clinics | 1 day
  Transition protocols will be assessed by one-time interviews with AMTU Clinic staff where youth from AMTUs transition their care within one year of site registration.
Transition Processes at AMTUs and Adult Clinics | 1 day
  Transition processes will be assessed by one-time interviews with AMTU Clinic staff where youth from AMTUs transition their care within one year of site registration.
Preparedness of Adult Clinics to Receive Behaviorally-Infected HIV-Positive Youth Transitioning from Adolescent Clinics | 1 day
  Preparedness will be assessed by one-time interviews with Adult Clinic staff where youth from AMTUs transition their care within one year of site registration.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Tanner, PhD, MPH, Study Chair — University of North Carolina, Greensboro; J. Dennis Fortenberry, MD, MS, Study Chair — Indiana University School of Medicine
Locations (14):
- United States (14):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of Colorado - The Children's Hospital of Denver, Aurora, Colorado
  - Children's Hosp Natinal Med Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: ATN Website — http://www.atnonline.org